CLINICAL TRIAL: NCT04150731
Title: 16α-18F-fluor-17β-østradiol PET/CT Til Visualisering af østrogenreceptor-positive Levermetastaser Fra brystkræft
Brief Title: 16α-18F-fluor-17β-estradiol PET/CT for Visualisation of Estrogen Receptor Positive Liver Metastases From Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); REDCap (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020FES
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Liver metastases; FES-PET/CT; Dynamic scan
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer and FES (Experimental): Only one arm: All included are patients with disseminated breast cancer and all have an experimental FES-PET/CT done
  Interventions: Radiation: 16α-18F-fluor-17β-estradiol

INTERVENTIONS:
Radiation: 16α-18F-fluor-17β-estradiol — 16α-18F-fluor-17β-estradiol PET/CT scan

SUMMARY:
Breast cancer (BC) is the most common cancer diagnosis among women and the incidence is increasing. Prognosis and treatment are dependent on the expression of estrogen receptors (ER) in the tumor. ER status is determined by immunohistochemistry (IHC) on biopsy tissue. The ER expression can change over time and be heterogeneous.

The IHC score on ER expression is subjective and can lead to intra and inter observer variability. A new computer image analysis software that can give the exact percentage of colored tumor cells on sectional tumor cuts has been developed.

It is also possible to quantify the ER expression non invasive by using the tracer 16α-18F-flour-17β-estradiol (FES) and in vivo positron emission tomography (PET) scans. FES-PET/CT has a high background activity in the liver which complicates the visualization of liver metastases. Theoretically, a new whole body parametric scan method makes it possible to distinguish background activity from uptake in liver metastases.

Malignant tumors often have an increased perfusion, and previous studies have found that tumors with low metabolism relative to blood flow have the longest disease free survival (DFS). To the best of our knowledge, no previous studies have examined the correlation between ER expression and blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known disseminated breast cancer
* Metastatic ER+ HER2- breast cancer with metastases in the liver, at least two separate liver foci visualised on CT
* Diagnostic CT scan done in connection with clinical control
* Treatment with aromatase inhibitors, and potential additional treatment
* Postmenopausal

Exclusion Criteria:

* Treatment with Tamoxifen or Fulvestrant completed within 5 weeks prior to FES-PET/CT
* ER- metastases
* Life expectancy under three months
* Claustrophobia
* Any pain which makes it impossible to lie in the scanner for 90 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity of parametric FES-PET/CT | 1 year
  Examine the sensitivity of parametric FES-PET/CT compared to conventional FES-PET/CT to detect estrogen receptor (ER) positive liver metastases

SECONDARY OUTCOMES:
Correlation of ER expression | 1 year
  Correlate the ER expression in metastases measured by parametric FES-PET/CT to Visiopharm H-score on biopsy material examined by immunohistochemistry (IHC)
Examination of the heterogeneity of ER expression in liver metastases | 1 year
  Examine intra-individual heterogeneity of ER expression in liver metastases by FES-PET/CT
Examination of the heterogeneity of ER expression i metastases | 1 year
  Examine intra-individual heterogeneity of ER expression in metastases in different tissues by FES-PET/CT
Examination of the heterogeneity of ER expression | 1 year
  Examine the heterogeneity of the ER expression between primary tumor and metastases by FES-PET/CT
Correlation of tumor blood flow to ER+ cells | 1 year
  Correlate tumor blood flow measured by H215O-PET/CT to the percentage of ER+ cells, measured by both FES-PET/CT and Visiopharm technology

CONTACTS AND LOCATIONS:
Overall Officials: Mette A Pedersen, MD, Principal Investigator — Department of Nuclear Medicine & PET-centre. Aarhus University Hospital, Denmark
Locations (1):
- Department of Nuclear Medicine & PET Centre, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen MA, Munk OL, Dias AH, Steffensen JH, Moller AL, Johnsson AL, Hansen KV, Bender D, Jakobsen S, Busk M, Gormsen LC, Tramm T, Borgquist S, Vendelbo MH. Dynamic whole-body [18F]FES PET/CT increases lesion visibility in patients with metastatic breast cancer. EJNMMI Res. 2024 Mar 4;14(1):24. doi: 10.1186/s13550-024-01080-y. PMID 38436824